CLINICAL TRIAL: NCT02767947
Title: A Randomized, Multi-Center, Double-Blind, Vehicle-Controlled Study Evaluating the Safety and Efficacy of Product 33525 in Pediatric Subjects With Tinea Corporis
Brief Title: Safety and Efficacy of Product 33525 (Luliconazole Cream 1%) in Pediatric Participants With Tinea Corporis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V01-LUZB-401; NCT02491112 (obsolete NCT alias)
Record Dates: First submitted 2016-05-06; First posted 2016-05-11 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Tinea Corporis
MeSH Terms: conditions — Tinea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Luliconazole Cream 1% (Experimental): Luliconazole cream 1% will be applied once daily in the morning for 7 days to the area affected with tinea corporis and approximately 1 inch of the immediate surrounding area.
  Interventions: Drug: Luliconazole Cream 1%
- Vehicle Cream (Placebo Comparator): Vehicle cream (containing no active ingredient) will be applied once daily in the morning for 7 days to the area affected with tinea corporis and approximately 1 inch of the immediate surrounding area.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: Luliconazole Cream 1% — Luliconazole cream will be applied per schedule specified in the arm.
  Other Names: Product 33525
  Arms: Luliconazole Cream 1%
Drug: Vehicle Cream — Vehicle cream will be applied per schedule specified in the arm.
  Arms: Vehicle Cream

SUMMARY:
The objective of this study was to evaluate the safety, efficacy, and pharmacokinetics of luliconazole cream 1% when applied topically for 7 days in pediatric participants 2 years to 17 years of age (inclusive) with tinea corporis.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants (or legal guardian/caregiver) with the ability and willingness to sign a written informed consent and/or assent (age appropriate).
* Participants of either gender must be at least 2 years to less than (<) 18 years of age (2 to 17 years, inclusive).
* Participants with a clinical diagnosis of tinea corporis characterized by clinical evidence of a tinea infection (at least moderate erythema, mild scaling, and moderate pruritus).
* Participants must be in good general health and free of any disease that in the Investigator's opinion might interfere with the study evaluations.
* Participants/caregiver must be able to communicate, be able to understand the study procedures, and be willing to comply with the study requirements.

Key Exclusion Criteria:

* Participants with active atopic or contact dermatitis in the area to be treated.
* Participants with severe dermatophytoses, mucocutaneous candidiasis, or bacterial skin infection.
* Female participants who are pregnant and/or nursing or planning a pregnancy during the course of the trial. Participants who test positive for pregnancy after start study drug will be discontinued from study drug but will be followed for safety purposes.
* Participants who are immunocompromised (due to disease, for example; human immunodeficiency virus [HIV] or medications).
* Participants who have a recent history of or current drug or alcohol abuse.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2016-02-08 (Actual); Primary Completion 2016-06-29 (Actual); Study Completion 2016-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Valeant Pharmaceuticals
Locations (3):
- Dominican Republic (2):
  - Valeant Site 03, San Cristóbal
  - Valeant Site 01, Santo Domingo
- Valeant Site 02, San Pedro Sula, Honduras

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 75 participants with tinea corporis were enrolled and randomized in 4:1 ratio to receive either luliconazole cream 1% or vehicle cream.
Groups:
- Luliconazole Cream 1%: Luliconazole cream 1% was applied once daily in the morning for 7 days to the area affected with tinea corporis and approximately 1 inch of the immediate surrounding area.
- Vehicle Cream: Vehicle cream (containing no active ingredient) was applied once daily in the morning for 7 days to the area affected with tinea corporis and approximately 1 inch of the immediate surrounding area.
Period: Overall Study
Arm/Group | Luliconazole Cream 1% | Vehicle Cream
Started | 60 | 15
Safety Population (Received at least 1 application of study drug.) | 60 | 15
Pharmacokinetic (PK) Population (Received at least 1 dose of study drug, and had blood samples obtained both pre and 6 hrs post-dose.) | 12 | 3
Completed | 60 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 application of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Luliconazole Cream 1% | Vehicle Cream | Total
Number analyzed (Participants) | 60 | 15 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.18 (3.87) | 9.13 (5.18) | 8.37 (4.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 3 | 21
  Male | 42 | 12 | 54

OUTCOME MEASURES:

1. Primary Outcome: Circulating Plasma Concentration of Luliconazole at Day 7 (Pre-Dose)
Description: Plasma levels of luliconazole were obtained at steady-state (within 15 minutes prior to the final dose of the study drug on Day 7) and approximately the time of maximum concentration (tmax) (6 hours after the final dose of study drug on Day 7).
Time Frame: Pre-dose (within 15 minutes prior to the final dose of the drug) on Day 7
Population: PK population included all randomized participants who received at least 1 application of study drug, and from whom blood samples were obtained for plasma level analysis both prior to (within 15 minutes) and 6 hours after the final dose (on Day 7).
Measure: Mean (Standard Deviation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Luliconazole Cream 1% | Vehicle Cream
Number analyzed (Participants) | 12 | 3
nanograms/milliliter (ng/mL) | 4.63 (2.93) | NA (NA) — Data not available due to concentration below the limit of quantitation.

2. Primary Outcome: Circulating Plasma Concentration of Luliconazole at Day 7 (6 Hours Post-Dose)
Description: Plasma levels of luliconazole were obtained at steady-state (within 15 minutes prior to the final dose of the study drug on Day 7) and approximately the tmax (6 hours after the final dose of study drug on Day 7).
Time Frame: 6 hours after the final dose of the drug on Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Luliconazole Cream 1% | Vehicle Cream
Number analyzed (Participants) | 12 | 3
ng/mL | 4.84 (3.33) | 0.07 (0.12)

ADVERSE EVENTS:
Time Frame: From Baseline (Day 1) to Day 28
Description: Safety population included all randomized participants who received at least 1 application of study drug.
Arm/Group | Luliconazole Cream 1% | Vehicle Cream
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/15
Other Adverse Events (participants affected / at risk) | 7/60 | 2/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Luliconazole Cream 1% (N=60) | Vehicle Cream (N=15)
Nasopharyngitis (Infections and infestations) | 4 | 2
Headache (Nervous system disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.